CLINICAL TRIAL: NCT04718129
Title: Targeting Negative Affect Through Mindfulness Training in Youth at Risk for Internalizing Problems - R61
Brief Title: Testing the Effect of the Youth Mindful Awareness Program on Negative Affect
Acronym: YMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Northwestern University (Other); University of California, Los Angeles (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Judith Garber, Principal Investigator, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 570035; R61MH119270 (NIH); R33MH119270 (NIH)
Record Dates: First submitted 2020-11-29; First posted 2021-01-22 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Mindfulness
Keywords: Mindfulness

STUDY DESIGN:
Intervention Model Description: Mindfulness vs. No intervention control
Who Masked: Outcomes Assessor
Masking Description: Assessors of outcomes will be masked to intervention condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): Internet-based, coached Mindfulness Program. Nine weekly coached sessions with practice exercises between sessions.
  Interventions: Behavioral: Youth Mindful Awareness Program (YMAP)
- Control (No Intervention): Participants in this arm are randomly assigned to an assessment-only, no intervention control condition.

INTERVENTIONS:
Behavioral: Youth Mindful Awareness Program (YMAP) — The Mindfulness Intervention is an internet-based program that involves a coach. It is 9 weekly sessions and involves practicing the skills between sessions.
  Arms: Mindfulness

SUMMARY:
Randomized controlled trial comparing a coached, app-based mindfulness intervention versus a no-intervention control condition. Primary outcome: adolescents' reports of affect as measured with ecological momentary assessment (EMA) at post-intervention. Participants will include 120 youth ages 12-17 years old.

DETAILED DESCRIPTION:
This is a randomized controlled trial testing a 9-session, coached, app-based mindfulness intervention on adolescents' reports of affect as measured with ecological momentary assessment (EMA). Participants will include 120 youth ages 12- to 17-years-old randomized to either the Youth Mindful Awareness Program (YMAP) or to an assessment only control condition. Participation is open to all genders and youth of all races and ethnicities.

ELIGIBILITY:
Inclusion Criteria:

* ages 12- to 17-years-old
* has access to a smartphone, tablet, or other mobile device on which they can access the mindfulness app and complete EMA reports. Youth without a device will be provided with one for their time in the study.

Exclusion Criteria:

* current DSM5 diagnosis of an anxiety or depressive disorder with significant clinical impairment
* current alcohol or substance use disorder; currently suicidal
* lifetime diagnosis of bipolar disorder, schizophrenia, autism, conduct disorder, or developmental delay
* reading level below 4th grade
* not English speaking at a level that would allow them to participate in the intervention and assessments.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy Garber, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Judy Garber, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Results will be shared through Clinical Trials.gov, and by the study PIs at scientific conferences and publications in scientific journals. IPD will be available upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after study completion and publications of study results.
Access Criteria: Access to study data will require a written request to the PIs. The request should include a description of the research question(s), planned analyses, and data requested.

REFERENCES:
- [Derived] Garber J, Chavira DA, Adam EK, Craske MG, McMahon T, Williams A, Abitante G, Lanser I, Pashtunyar DS, Chen S, Zinbarg R. A randomized controlled trial of an online mindfulness program for adolescents at risk for internalizing problems. J Consult Clin Psychol. 2025 Apr;93(4):226-237. doi: 10.1037/ccp0000921. Epub 2024 Dec 2. PMID 39621373

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through a university listserv, advertising on FaceBook and in subways (in Chicago), local schools, and community events. Recruitment began 05/15/2021
Pre-assignment Details: After parents completed the consent form and the teen completed the assent form, the teen was interviewed regarding the inclusion and exclusion criteria (e.g., psychiatric symptoms and diagnoses).
Period: Overall Study
Arm/Group | Mindfulness | Control
Started | 53 | 57
Completed | 47 (Analyses were "intent to treat" and conducted on all 53 participants randomized to this condition.) | 50 (Seven participants discontinued participation. Analyses were "intent to treat" and included all 57 participants in this condition.)
Not Completed | 6 | 7
Not completed — Lost to Follow-up | 6 | 7

BASELINE CHARACTERISTICS:
Population: All 110 randomized participants were included in the "intent to treat" analyses regardless of attrition.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness | Control | Total
Number analyzed (Participants) | 53 | 57 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.13 (1.68) | 14.20 (1.53) | 14.17 (1.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 40 | 76
  Male | 17 | 17 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 16 | 36
  Not Hispanic or Latino | 33 | 41 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 33 | 35 | 68
  More than one race | 10 | 14 | 24
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 57 | 110

OUTCOME MEASURES:

1. Primary Outcome: Momentary Negative Affect Assessed With Ecological Momentary Assessment
Description: Momentary negative affect (mNA) in EMA is the experience of negative emotional states in the moment. Participants complete the Ecological Momentary Assessment (EMA) 4 times a day for 5 days, at random moments across the day (usually once in the morning, once in the early afternoon, once in the late afternoon and once in the evening). The EMA affect measure includes 7 items rated on a 4-point scale; average scores range from 1.00 to 4.00; higher scores indicate more negative affect (NA).
Time Frame: 5 days
Population: All 110 randomized participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness | Control
Number analyzed (Participants) | 53 | 57
score on a scale | -.17 (1.39) | .14 (.25)
Statistical Analysis 1: Comparison: Mindfulness vs Control; Test type: Superiority; p = .048, Regression, Linear; Mean Difference (Net) = .044, 95% CI 2-sided [.003 to .085], Standard Error of Mean .021

ADVERSE EVENTS:
Time Frame: Two years
Description: The definition of adverse event and serious adverse event used to collect adverse event information was from the clinicaltrials.gov Definitions.
Groups:
- Control: Participants in this arm were randomly assigned to an assessment-only, no intervention control condition.
Arm/Group | Mindfulness | Control
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/57
Other Adverse Events (participants affected / at risk) | 0/53 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT04718129/Prot_002.pdf
  • Statistical Analysis Plan (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT04718129/SAP_003.pdf
  • Informed Consent Form: ICF parent part 2 (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/29/NCT04718129/ICF_000.pdf
  • Informed Consent Form: ICF parent part 1 (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/29/NCT04718129/ICF_001.pdf